CLINICAL TRIAL: NCT06306586
Title: Evaluation of a Personalised Digital Treatment for Adolescents With Eating Disorders - An Open Feasibility Trial in Routine Care
Brief Title: A Digital Treatment for Adolescents With Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Fonna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 639031
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders
Keywords: Digital interventions, eating disorders, adolescents
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Treatment for Adolescents With Eating Disorders (Experimental): The digital treatment is guided by a therapist and comprises 8 modules, running over a span of 10 weeks.
  Interventions: Behavioral: Digital Treatment for Adolescents With Eating Disorders

INTERVENTIONS:
Behavioral: Digital Treatment for Adolescents With Eating Disorders — The main aim of the digital treatment is to reduce symptoms of eating disorders and increase life-coping skills. The digital treatment aims to help adolescents with eating disorders to:
  * Gain knowledge about the symptoms of eating disorders and the consequences it has on everyday life.
  * Be motivated to carry out the treatment.
  * Gain knowledge of and skills in regulating food and activity in a more balanced way.
  * Gain knowledge of and skills in managing emotions.
  * Get tools to develop a better self-esteem.
  * Gain awareness of the function of the eating disorder.
  * Gain skills in coping with social challenges.
  * Get a more realistic image of their bodies and handle information from social media.
  Other Names: e-balanse

SUMMARY:
The goal of this feasibility study is to evaluate the feasibility and preliminary clinical outcomes of a personalized digital treatment for adolescents with eating disorders. The main objectives are to:

i) Evaluate whether a personalized digital treatment for adolescents with eating disorders are feasible in a child and adolescent psychiatric outpatient clinic.

ii) Evaluate who benefits from a personalized digital treatment for adolescents with eating disorders (what works for whom?) iii) Evaluate the cost-benefit of a personalized digital treatment for adolescents with eating disorders.

Participants will be enrolled in a 10-week digital treatment including weekly therapist contact. They will be asked to complete self-report questionnaires at pre-, during, post- and 3- and 6-months follow-up.

DETAILED DESCRIPTION:
Eating disorders are associated with high levels of distress, significant somatic problems, and high mortality. The difficulties have significant consequences for the individual, family members, and society at large. Early treatment leads to better prognosis, but the identification and treatment of eating disorders are challenging within the healthcare system. The effect of digital treatments for patients with eating disorders appears promising.

In this study, we will investigate the feasibility and preliminary effects of therapist-guided digital treatment for youth with eating disorders using qualitative and quantitative methods. The project uses the Person-based approach (PBA) as methodological framework, which is an evidence-based method for developing user-centered and effective behavior change interventions.

The study wants the examine the intervention within six feasibility domains that includes the following research questions:

Feasibility domain 1. Sample distribution of general psychopathology of eating disorder symptoms:

A. Will a reasonable wide spectrum of individuals with different forms of eating disorders show interest and be eligible? B. Will 60 adolescents be eligible over the course of one year? C. What characterizes the group that participate (predictor)?

Feasibility domain 2. Adherence to the treatment protocol:

A. Do 50% of the adolescents complete the entire intervention? B, What characterizes those who carry out the treatment (predictor)? C. What characterizes those who drop out (predictor)?

Feasibility domain 3. Treatment credibility:

A. Will 70% of the participants rate the treatment as acceptable/recommend it to a friend?

Feasibility domain 4. Treatment acceptability:

A. What are the adolescents' experiences of a personalised digital treatment targeting eating disorders?

Feasibility domain 5. Treatment use and utility:

A. Will a moderate within-group effect, around d=0.50, be seen on general psychopathology of eating disorder? B. Will more than 40% of the sample obtain a significant reliable change on primary outcome? C. Will less than 10% of the sample experience negative effects and/or deterioration defined as a negative significant reliable change?

Feasibility domain 6. Treatment cost-effectiveness:

A. What is the cost-effectiveness of a personalized digital treatment for for adolescents with eating disorders in routine care?

Youth between the ages of 16-18 with an eating disorder will be invited to participate in this intervention study. The participants will be recruited via child and youth psychiatric outpatient clinics and social and media. Eligible participants get access to an online information consent form which is signed digitally using the Norwegian electronic identification system BankID.

Data will be collected using self-report questionnaires administrated online at pre-, during, post- and 3- and 6-months follow-up. All measures are previously validated and have been used in eating disorder adolescent populations. Based on the literature potential predictors are included in the study protocol. The pre-treatment symptoms variables are associated with external clinical features, which maintain an eating disorder. The predictor variables will be collected pre-treatment.

We will conduct semi-structured phone interviews to explore the patients' in-depth experience of the digital treatment. The interviews of approximately 16 adolescents will be conducted 2-4 weeks after finishing the treatment. We will strive to have two groups, one with participants that finished the treatment, and one with dropouts.

ELIGIBILITY:
Inclusion Criteria:

A. Diagnosed with F50.1 Atypical anorexia nervosa, F50.3 Atypical bulimia nervosa, F50.8 Other eating disorders, F50.9 Eating disorder, unspecified

B. Age between 15 and 18 years.

C. Stable dose of medication for a co-morbid psychiatric treatment for six weeks and who continue to meet study entry criteria.

D. Internet access.

E. Speaks and write Norwegian.

Exclusion Criteria:

A. Diagnosed with F50.0 Anorexia nervosa or F50.2 Bulimia nervosa

B. Disorders of psychological development (F80-F89).

C. Patients with avoidant restrictive food intake disorders (F50.82)

D. Participants with a co-morbid medical condition or disorder known to influence eating or weight (i.e., pregnancy, cancer), psychotic disorders, acute suicidality, or substance abuse and/or substance dependence and severe depressive episode.

E. Receiving inpatient- or face to face psychological treatment.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The Credibility and Expectancy Scale (CEQ-1) | One week
  CEQ-1 will be used after participants have completed the first module of the treatment. CEQ measures perceived treatments credibility. We will use 1-item "How confident would you be in recommending this treatment to a friend who experiences similar problems?" The item is rated on a scale from 0 to 10, where higher score indicates better treatment credibility.
Adherence | Up to 10 weeks
  Adherence (dropout rates and completion of modules) will be used to assess the acceptability of the intervention. The total number of logged on sessions during the intervention period will be collected, and the average length of sessions. Days in treatment will be calculated based on the dates between the first login, and the completion of the last module.
Module evaluations | Up to 10 weeks
  After each treatment module the participants will be asked to evaluate the module which will be used to assess acceptability of the intervention. With a 6-item self-report questionnaire assessed on a 5-point Likert scale ranging from "completely disagree" to "completely agree".
Client Satisfaction Questionnaire (CSQ-3) | 10 weeks
  Intervention satisfaction will be measured at post-treatment, using the 3-item Client Satisfaction Questionnaire (CSQ-3) CSQ-3 are items 3, 7, & 8 from the CSQ-8. Each item on the CSQ-3 is scored from 1 to 4, where a higher score indicate higher satisfaction.
Recruitment | 1 year
  Number of participants of participants recruited and inclusion rate will be used to assess the acceptability.
Eating disorder symptoms | Up to 6-months follow-up
  Eating Disorder Examination-Questionnaire Short (EDE-QS) is a 12 item self-report questionnaire that with a 4-point response scale assess eating disorder symptom severity over the preceding 7 days. It has demonstrated good psychometric properties at initial testing.
The Clinical Impairment Assessment Questionnaire (CIA) | Up to 6-months follow-up
  We will use the The Clinical Impairment Assessment Questionnaire (CIA) to assess quality of life. CIA assess the severity of psychosocial impairment due to eating disorder features. It is a 16-item self-report questionnaire that cover impairment in domains of life that are typically affected by eating disorder psychopathology: mode and self-perception, cognitive functioning, interpersonal functioning, and work performance.
The KIDSCREEN (KIDSCREEN-10) | Up to 6 months follow-up
  The KIDSCREEN (KIDSCREEN-10) will be used to assess quality of life. The items are rated on 5-point Likert scale that indicates the frequency or intensity of a behavior or emotion.

SECONDARY OUTCOMES:
The Patient Health Questionnaire (PHQ-2) | Up to 6-months follow-up
  The Patient Health Questionnaire (PHQ-2) are used for assessing depression. The PHQ-2, comprising the first 2 items of the PHQ-9, inquiries about the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks. Items are rated on scale from 1 to 4, where a higher rating indicate higher degree of depressed mood.
Generalized Anxiety Disorder scale (GAD-2) | Up to 6-months follow-up
  Generalized Anxiety Disorder scale (GAD-2) is used for assessing anxiety disorders. The GAD-2 is a quick version of the seven-item scale that incorporates the first two questions of the GAD-7, which are also critical components of any anxiety disorder.Items are rated on scale from 1 to 4, where a higher rating indicate higher degree of anxiety.
School attendance | Up to 6-months follow-up
  In addition, we will collect School attendance (variables: full-time/reduce-time/don't attend school/ don't attend school but have a job) to assess quality of life.
Tme with friends | Up to 6-months follow-up
  Time with friends with the categories: daily/weekly/monthly/don't have friends/ don't have time to friends because of my eating disorder, will also be used to assess quality of life.
Difficulties with Emotion Regulation Scale (DERS-18) | Up to 6-months follow-up
  Difficulties with Emotion Regulation Scale (DERS-18) are used to assess used to facilitate understanding of how emotion dysregulation is associated with psychiatric symptoms, other emotion-related constructs, and treatment progress. Responses are rated one a scale from 1 to 5, ranging from never to almost always, where a higher score indicates higher severity.
EuroQoL 5D-5L (EQ-5D-5L) | Up to 6-months follow-up
  EuroQoL 5D-5L (EQ-5D-5L) measures health-related quality of life and provide data for calculation of Quality Adjusted Life Years (QALY), to be used in the economic evaluation. The questionnaire covers five dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), identify the health states and together with preference scores provides a single index score in order to calculate QALYs.

OTHER OUTCOMES:
The Rosenberg Self-Esteem Scale (RSES) | Baseline
  The Rosenberg Self-Esteem Scale (RSES) to measure self-esteem, a maintaining mechanism. RSES is a widely used 10-item self-report questionnaire. Items are answered on a 4-point scale, ranging from 3 (strongly agree) to 0 (strongly disagree). Scores range from 0 to 40, and higher scores indicate higher global self-worth.
The readiness to change questionnaire (RTCQ-6) | Baseline
  The readiness to change questionnaire (RTCQ-6) is adapted to the study population and digital treatment inspired by the Short Motivation Feedback List (SMFL-8).
Qualitative interviews | Up to 4 weeks post-treatment
  Qualitative interviews will be conducted following the intervention with 16 participants. We will aim to recruit both treatment completers and treatment dropouts.

CONTACTS AND LOCATIONS:
Overall Officials: Tine Nordgreen, PhD, Principal Investigator — Division of Psychiatry, Haukeland University Hospital
Locations (3):
- Norway (3):
  - Bømlo Kommune, Bømlo, Vestland
  - Haukeland University Hospital, Bergen
  - Helse Fonna, Haugesund